CLINICAL TRIAL: NCT04976049
Title: Use of 5-Aminolevulinic Acid to Assess Bone and Tissue Profusion in Orthopaedic Infection Patients
Status: Withdrawn | Type: Observational
Why Stopped: Principle Investigator decided not to pursue study
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Associate Professor of Orthopaedics, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02000990
Record Dates: First submitted 2021-06-02; First posted 2021-07-26 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Trauma; Infection; Bone Fracture
Keywords: 5-Aminolevulinic Acid, infection, orthopedics, imaging
MeSH Terms: conditions — Wounds and Injuries; Infections; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic infection: Subjects who have undergone previous trauma surgeries and have developed an infection will be assessed for protocol inclusion criteria. Patients will be administered a single, oral, 20mg/kg dose of 5-Aminolevulinic Acid (ALA) by a qualified member of their care team. This dose will be administered ideally 3 hours prior to surgery. Fluorescent imaging will be obtained pre and post irrigation and debridement.
  Interventions: Procedure: Imaging using 5-Aminolevulinic Acid (5-ALA) during surgery

INTERVENTIONS:
Procedure: Imaging using 5-Aminolevulinic Acid (5-ALA) during surgery — Patients will be administered FDA approved oral 5-ALA and imaged by a FDA approved surgical fluorescence imaging device (Spy Elite) which is 0.5 meter away from the subject.

SUMMARY:
The focus of this study is to explore the variability distribution of 5-Aminolevulinic Acid (ALA)associated with bone and soft tissue perfusion in infection patients, using 5-ALA fluorescence imaging. In additional this study plans to evaluate the change in 5-ALA distribution from pre to post debridement and to preliminarily determine whether an orally administered dose of 20mg/kg 5-ALA can predict recurrent infection/treatment failure.

DETAILED DESCRIPTION:
The focus of this study is to (1) Explore variability in distribution of 5-Aminolevulinic Acid (ALA) in bone and soft tissue infection (2) Evaluate the change in 5-ALA distribution from pre to post debridement (3) Preliminarily determine whether 5-ALA has the possibility predict infection / treatment failure

Infection following trauma is one of the most prevalent and challenging complications faced by orthopedic surgeons in both military and civilian populations, occurring after up to 60% of open bone fractures. Several factors specific to this trauma place patients at high risk for infectious complications, including: traumatized tissues, open contaminated fracture, soft tissue coverage issues, catabolic state due to poly-trauma, prolonged hospitalization with exposure to nosocomial bacteria, and presence of metallic implants8. Infection requires one or more unplanned surgical procedures and leads to prolonged morbidity, loss of function, and potential loss of limb1. Failed treatment for bone infection results in recurrent infection, requiring repeat surgical procedures in approximately 30% of patients.

Studies are currently being conducted to evaluate the utility of first window Indocyanine Green (ICG) to identify areas of deficient perfusion. This is based upon the concept deficient perfusion prevents delivery of antibiotics and endogenous immune cells to traumatized tissues. In the setting of established infection, poorly perfused bone can be a nidus for biofilm formation creating resistance to antibiotics. However, in the context of this work it is becoming increasingly clear that acute (rather than chronic) infections display hyper vascularity with increased blood flow and neovascularization. Infection is known to display the enhanced permeability and retention effect with increased vascular permeability.

There are currently no accepted intraoperative tools that can be used to make objective decisions about which bone and tissue is infected and which is normal. Methods currently used to guide debridement are quite rudimentary. Clinical judgement is based on the gross appearance of soft tissue and bone, including color, turgor, and extent of soft tissue stripping. A burr may be used to look for bleeding bone. More extensive debridement is thought to minimize risk of index infection or reduce the rate of persistent infection; however, this comes at the cost of increasingly complex reconstructive procedures to fill bony defects. Clearly what is needed is a functional imaging system which can identify infected tissues to guide surgeons in the amount of tissue to debride. In turn, this will lead to fewer infections and a more effective treatment of surgical site infections (SSIs) at the fracture site. Both scenarios will allow patients to return to duty or work sooner.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older.
2. History of an extremity fracture.
3. Prior definitive fracture management with external fixation, internal fixation, or joint fusion.
4. Superficial, deep, or organ space surgical site infection (SSI) (as per Center for Disease Control criteria) at the fracture site that requires operative management.
5. Will have all planned SSI care surgeries performed by a participating surgeon or delegate.
6. Provision of informed consent.

Exclusion Criteria:

1. Fractures of the hand cannot be imaged.
2. Iodine allergy.
3. Burns at the SSI site.
4. Incarceration.
5. Expected survival of less than 90 days.
6. Problems, in the judgment of study personnel, with maintaining follow-up with the patient.
7. Adults unable to consent or whom do not have a legal authorized representative
8. Individuals who are not yet adults (infants, children, teenagers)
9. Pregnant or breastfeeding women
10. History of cutaneous photosensitivity, porphyria, hypersensitivity to porphyrins, photodermatosis, exfoliative dermatitis.
11. History of liver disease within the last 12 months.
12. Elevated liver function tests (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase or bilirubin levels greater than 2.5 times the normal limit) from laboratory tests conducted within 30 days prior to surgery.
13. Serum creatinine in excess of 180 µmol/L within 30 days prior to surgery.
14. Inability to comply with the photosensitivity precautions associated with the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who present to Dartmouth-Hitchcock Medical Center with an orthopaedic infection
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
5-Aminolevulinic Acid distribution variability | One Day
  Distribution of 5-Aminolevulinic Acid in the bone and soft tissue of infection patients, measured using fluorescent imaging.

SECONDARY OUTCOMES:
5-Aminolevulinic Acid distribution pre and post debridement. | One Day
  Distribution of 5-Aminolevulinic Acid in bone and soft tissue prior to and following debridement, measure using fluorescent imaging

OTHER OUTCOMES:
5-Aminolevulinic Acid Dose Effectiveness | 6 months
  Number of patients who do not experience a recurrent infection following the experimental dose of 5-Aminolevulinic Acid.

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No